CLINICAL TRIAL: NCT06962878
Title: Assessment of Bone Volume Changes in Immediate Implant Placement Using Allograft Versus Xenograft in Mandibular Molars: Randomized Clinical Trial
Brief Title: Assessment of Bone Volume Changes in Immediate Implant Placement Using Allograft Versus Xenograft in Mandibular Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Tawfik, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Grafting in immediate implants
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-05

CONDITIONS: Bone Volume; Immediate Implant With Bone Graft
Keywords: Bone graft; Jumping gap; Xenograft; Allograft; Immediate implant
MeSH Terms: interventions — Transplantation, Heterologous; Transplantation, Homologous

STUDY DESIGN:
Who Masked: Participant
Masking Description: This trial is considered a randomized single blind clinical trial due to the following:
  * The participants will be blinded to the technique that will be used during the surgical procedure.
  * The operator will not be blinded for both techniques during the surgical procedure as the two techniques are different.
  * The outcome assessor cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xenograft (Active Comparator)
  Interventions: Procedure: Xenograft
- Allograft (Experimental)
  Interventions: Procedure: Allograft

INTERVENTIONS:
Procedure: Xenograft — The jumping gap and surrounding space will be augmented and packed with Xenograft
  Arms: Xenograft
Procedure: Allograft — The jumping gap and surrounding space will be augmented and packed with Allograft
  Arms: Allograft

SUMMARY:
Twenty recruited patients indicated for immediate implant placement in mandibular molar sites are divided into two groups, with each group containing ten patients. One group assigned for placement of xenograft after molar extraction and immediate implant placement, while the other group received allograft as space-filling material.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-restorable mandibular molars
* Both sexes with age range from 25 years to 40 years
* Good oral hygiene
* Adequate alveolar bone dimensions for implant replacement
* Adequate bone volume after extraction to achieve primary stability of the immediate implant
* Co-operative patient

Exclusion Criteria:

* Patients with any systemic disease as uncontrolled diabetes or osteoporosis
* Heavy smokers with smokers more than 10 cigarettes per day
* Pregnancy
* Patients with any signs of active infection or pus formation
* Patients undergoing chemotherapy or radiotherapy, immunocompromised patients

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone thickness in millimeters | 6 months postoperative
  Two CBCT images will be taken, one immediately after surgery (baseline) and the other at 6 months post-surgically

SECONDARY OUTCOMES:
Vertical bone height in millimeters | 6 months postoperative
  Two CBCT images will be taken, one 2 days after surgery (baseline) and the other at 6 months post-surgically
Pain intensity | One week postoperative
  The pain will be recorded by participants at 1, 3, and 7 days after surgery using the Visual Analogue Scale (VAS), which ranges from 0 to 10. The minimum score is 0, indicating no pain, and the maximum score is 10, representing the worst possible pain. Higher scores on the VAS indicate worse outcomes in terms of pain experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Atef, PhD, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Botticelli D, Berglundh T, Buser D, Lindhe J. The jumping distance revisited: An experimental study in the dog. Clin Oral Implants Res. 2003 Feb;14(1):35-42. doi: 10.1034/j.1600-0501.2003.140105.x. PMID 12562363
- [Background] Bhola M, Neely AL, Kolhatkar S. Immediate implant placement: clinical decisions, advantages, and disadvantages. J Prosthodont. 2008 Oct;17(7):576-81. doi: 10.1111/j.1532-849X.2008.00359.x. Epub 2008 Aug 26. PMID 18761580
- [Background] Lang NP, Pun L, Lau KY, Li KY, Wong MC. A systematic review on survival and success rates of implants placed immediately into fresh extraction sockets after at least 1 year. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:39-66. doi: 10.1111/j.1600-0501.2011.02372.x. PMID 22211305
- [Background] Dimitriou R, Mataliotakis GI, Angoules AG, Kanakaris NK, Giannoudis PV. Complications following autologous bone graft harvesting from the iliac crest and using the RIA: a systematic review. Injury. 2011 Sep;42 Suppl 2:S3-15. doi: 10.1016/j.injury.2011.06.015. Epub 2011 Jun 25. PMID 21704997
- [Background] Khoury F, Hanser T. Mandibular bone block harvesting from the retromolar region: a 10-year prospective clinical study. Int J Oral Maxillofac Implants. 2015 May-Jun;30(3):688-97. doi: 10.11607/jomi.4117. PMID 26009921
- [Background] Schropp L, Isidor F. Timing of implant placement relative to tooth extraction. J Oral Rehabil. 2008 Jan;35 Suppl 1:33-43. doi: 10.1111/j.1365-2842.2007.01827.x. PMID 18181932
- [Background] Alexopoulou M, Lambert F, Knafo B, Popelut A, Vandenberghe B, Finelle G. Immediate implant in the posterior region combined with alveolar ridge preservation and sealing socket abutment: A retrospective 3D radiographic analysis. Clin Implant Dent Relat Res. 2021 Feb;23(1):61-72. doi: 10.1111/cid.12974. Epub 2021 Jan 13. PMID 33438320
- [Background] Howe MS, Keys W, Richards D. Long-term (10-year) dental implant survival: A systematic review and sensitivity meta-analysis. J Dent. 2019 May;84:9-21. doi: 10.1016/j.jdent.2019.03.008. Epub 2019 Mar 20. PMID 30904559
- [Background] Adell R, Lekholm U, Rockler B, Branemark PI. A 15-year study of osseointegrated implants in the treatment of the edentulous jaw. Int J Oral Surg. 1981 Dec;10(6):387-416. doi: 10.1016/s0300-9785(81)80077-4. PMID 6809663
- [Background] Kononen E, Gursoy M, Gursoy UK. Periodontitis: A Multifaceted Disease of Tooth-Supporting Tissues. J Clin Med. 2019 Jul 31;8(8):1135. doi: 10.3390/jcm8081135. PMID 31370168
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31370168/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/6809663/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21704997/
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC5455762/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/1659621/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/356184/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22211305/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/16519184/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/18761580/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12562363/